CLINICAL TRIAL: NCT06764745
Title: Effect of Different Ventilation Modes on POCD in Elderly Patients with Abdominal Wall Hernia: a Randomized Controlled Trial
Brief Title: Effect of Different Ventilation Modes on POCD in Elderly Patients with Abdominal Wall Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inner Mongolia University of Science and Technology (Other)
Collaborators: Inner Mongolia Baogang Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other)
Responsible Party: Principal Investigator, Yu-Long Jia, Principal Investigator, Inner Mongolia University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MER-076
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Cognitive Impairment; Optic Nerve Sheath Edema
Keywords: Ventilation patterns; Elderly patients; Abdominal wall hernia; Postoperative cognitive impairment
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- PC Ventilation patterns Group (Experimental): Ventilation Modes Following induction, Group I patients received mechanical ventilation using the PC mode.
  Interventions: Device: PC Ventilation Modes
- VC Ventilation patterns Group (Experimental): Ventilation Modes Following induction, Group II patients received mechanical ventilation using the VC mode.
  Interventions: Device: VC Ventilation Modes
- PRVC Ventilation patterns Group (Experimental): Ventilation Modes Following induction, Group III patients received mechanical ventilation using the PRVC mode.
  Interventions: Device: PRVC Ventilation Modes

INTERVENTIONS:
Device: PC Ventilation Modes — Following induction, Group I patients received mechanical ventilation using the PC mode. The anesthetic machine (MAQUET Flow-I, Italy) parameters were set as follows: The inspiratory pressure (Pins) was adjusted to maintain an end-tidal carbon dioxide concentration (ETCO2) of 4.0-5.0 kPa. Pure oxygen and air were utilized at 0.3 L/min each, with an oxygen content of 41%. The positive end-expiratory pressure (PEEP) was set at 10 cmH2O, with an inspiration-to-expiration ratio of 1:2, a respiratory rate of 16 breaths per minute, and an oxygen content of 41%.
  Arms: PC Ventilation patterns Group
Device: VC Ventilation Modes — Following induction, Group II patients received mechanical ventilation using the VC mode. The anesthetic machine (MAQUET Flow-I, Italy) parameters were set as follows: The inspiratory pressure (Pins) was adjusted to maintain an end-tidal carbon dioxide concentration (ETCO2) of 4.0-5.0 kPa. Pure oxygen and air were utilized at 0.3 L/min each, with an oxygen content of 41%. The positive end-expiratory pressure (PEEP) was set at 10 cmH2O, with an inspiration-to-expiration ratio of 1:2, a respiratory rate of 16 breaths per minute, and an oxygen content of 41%.
  Arms: VC Ventilation patterns Group
Device: PRVC Ventilation Modes — Following induction, Group III patients received mechanical ventilation using the PRVC mode. The anesthetic machine (MAQUET Flow-I, Italy) parameters were set as follows: The inspiratory pressure (Pins) was adjusted to maintain an end-tidal carbon dioxide concentration (ETCO2) of 4.0-5.0 kPa. Pure oxygen and air were utilized at 0.3 L/min each, with an oxygen content of 41%. The positive end-expiratory pressure (PEEP) was set at 10 cmH2O, with an inspiration-to-expiration ratio of 1:2, a respiratory rate of 16 breaths per minute, and an oxygen content of 41%.
  Arms: PRVC Ventilation patterns Group

SUMMARY:
The purpose of this clinical trial is to understand the effect of different ventilation patterns during surgery on postoperative cognitive impairment in elderly patients with abdominal wall hernias. It will also explore how to reduce the incidence of postoperative cognitive impairment. The main questions it aims to answer are:

* Does the mode of ventilation affect the incidence of postoperative cognitive impairment in elderly patients?
* Does optic nerve sheath edema affect the incidence of postoperative cognitive impairment in elderly patients? Researchers will monitor patients with different ventilation patterns intraoperatively and investigate postoperatively to see if the ventilation pattern affects postoperative cognitive impairment.

Participants will:

* Randomly assigned to groups with different ventilation patterns
* Record various values during surgery by the researchers
* Presence of cognitive impairment assessed by cognitive scales after surgery

ELIGIBILITY:
Inclusion Criteria:

* Age: 65-90 years
* patients with abdominal wall hernias
* American Society of Anesthesiologists general status (ASA-PS) classes II and III.

Exclusion Criteria:

* Emergency (rather than elective) surgery or other types of surgery required
* More than one surgery required during hospitalization
* Preoperative demonstrated inability to communicate (due to coma, severe dementia, Parkinson's disease, severe hearing or visual impairment, or speech impairment).

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 471 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
MMSE scale | From enrollment to two weeks after surgical treatment
  Range Score <21 Increased odds of dementia Score >25 Decreased odds of dementia Education Score < 21 Abnormal for 8" grade Score <23 Abnormal for high school education Score <24 Abnormal for college education Severity 24-30 No cognitive impairment 18-23 Mild cognitive impairment 0-17 Severe cognitive impairment
optic nerve sheath diameter (ONSD) | From induction of anesthesia to the end of surgery
  The ONSD was assessed using ocular ultrasonography to non-invasively capture ICP. Bedside ultrasound measurements of the ONSD were performed by an experienced and professionally qualified ultrasound physician. Patients were positioned supine with their eyes softly closed, and their eyes were protected with disposable transparent patches. A 7.5 MHz linear probe (Micromaxx Ultrasound System; SonoSite Inc., Bothell, WA, USA) was gently placed on the closed upper eyelid without applying pressure to the eyeball, and sufficient ultrasound gel was applied to ensure clear imaging. The optic nerve sheath was checked and measured 3 mm beyond the globe, and three ONSD measures were performed, with the average value utilized as the final ONSD measurement, which was accurate to 0.01 mm.
average airway pressure( PAWM) | From induction of anesthesia to the end of surgery
  Mean airway pressure affects the patient's alveolar oxygenation status and blood circulation. Mean airway pressure is most affected by positive end-expiratory pressure, followed by prolongation of inspiratory time, which can also increase mean airway pressure.
esophagealp ressure（PES) | From induction of anesthesia to the end of surgery
  Esophageal pressure monitoring is a minimally invasive and clinically available method for estimating transpulmonary pressure, of which absolute values and changes are considered one of the main determinants of lung injury due to mechanical forces applied during mechanical ventilation . PES was monitored using a floating catheter (Swan-Ganz, USA) placed into the esophagus and coupled to a monitor (M8003A, Germany).
PaCO2(mmHg) | From induction of anesthesia to the end of surgery
  Arterial reference value: 35-45 mmHg, exceeding or falling below the reference value is called hyper- or hypocapnia. Exceeding 55mmHg may inhibit the respiratory center. It is the main index to determine the acid-base poisoning of each type.
mean arterial pressure（MAP） | From induction of anesthesia to the end of surgery
  Above 60 mmHg is sufficient to provide organ sustenance in the general population.calculated as MAP = diastolic pressure + 1/3 pulse pressure difference.
heart rate(HR） | From induction of anesthesia to the end of surgery
  Normal values for heart rate are 60-100 beats per minute.

SECONDARY OUTCOMES:
Aβ1-40 (pg·mL-1) | From induction of anesthesia to the end of surgery
  In the morning, 10 mL of venous blood from the upper limbs was withdrawn under fasting conditions, put into polypropylene EDTA anticoagulation tubes, centrifuged at 1 000 r/min for 3 min within 60 min (maximal centrifugal force: 27 700×g), and plasma was extracted, frozen in a refrigerator at -20 ℃, and then left to be measured. Plasma Aβ1-40 and inflammatory indexes were detected by enzyme-linked immunosorbent assay in the two groups.
S100 (pg·mL-1) | From induction of anesthesia to the end of surgery
  In the morning, 10 mL of venous blood from the upper limbs was withdrawn under fasting conditions, put into polypropylene EDTA anticoagulation tubes, centrifuged at 1 000 r/min for 3 min within 60 min (maximal centrifugal force: 27 700×g), and plasma was extracted, frozen in a refrigerator at -20 ℃, and then left to be measured. Plasma Aβ1-40 and inflammatory indexes were detected by enzyme-linked immunosorbent assay in the two groups.
IL-1β (pg·mL-1) | From induction of anesthesia to the end of surgery
  In the morning, 10 mL of venous blood from the upper limbs was withdrawn under fasting conditions, put into polypropylene EDTA anticoagulation tubes, centrifuged at 1 000 r/min for 3 min within 60 min (maximal centrifugal force: 27 700×g), and plasma was extracted, frozen in a refrigerator at -20 ℃, and then left to be measured. Plasma Aβ1-40 and inflammatory indexes were detected by enzyme-linked immunosorbent assay in the two groups.
IL-6 (pg·mL-1) | From induction of anesthesia to the end of surgery
  In the morning, 10 mL of venous blood from the upper limbs was withdrawn under fasting conditions, put into polypropylene EDTA anticoagulation tubes, centrifuged at 1 000 r/min for 3 min within 60 min (maximal centrifugal force: 27 700×g), and plasma was extracted, frozen in a refrigerator at -20 ℃, and then left to be measured. Plasma Aβ1-40 and inflammatory indexes were detected by enzyme-linked immunosorbent assay in the two groups.
TNF-α (pg·mL-1) | From induction of anesthesia to the end of surgery
  In the morning, 10 mL of venous blood from the upper limbs was withdrawn under fasting conditions, put into polypropylene EDTA anticoagulation tubes, centrifuged at 1 000 r/min for 3 min within 60 min (maximal centrifugal force: 27 700×g), and plasma was extracted, frozen in a refrigerator at -20 ℃, and then left to be measured. Plasma Aβ1-40 and inflammatory indexes were detected by enzyme-linked immunosorbent assay in the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baosteel Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Undecided